CLINICAL TRIAL: NCT03783611
Title: Testing the Effectiveness of MyPlan 2.0. on Physical Activity in Older Adults
Brief Title: Effectiveness of MyPlan 2.0. in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Principal Investigator, Vakgroepsport, Department of Movement and Sports Sciences, University Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MyPlan2.0._olderadults
Record Dates: First submitted 2018-12-12; First posted 2018-12-21 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Physical Activity; Older Adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group has access to the MyPlan 2.0. eHealth intervention. MyPlan is a eHealth intervention designed to increase physical activity. The intervention is based on the self-regulation theory and focuses on pre- and post-intentional processes to increase physical activity.
  Interventions: Behavioral: MyPlan 2.0.
- control group (No Intervention): The control group receives no intervention

INTERVENTIONS:
Behavioral: MyPlan 2.0. — eHealth intervention to increase physical activity in older adults. MyPlan 2.0 consists of five website visits. The first website visit contains pre- and post-intentional processes. The following four website visits contains mainly post-intentional processes. During the first website, participants fill in a questionnaire about their physical activity levels, and receive feedback. Furthermore, they are asked to make an action plan and think about barriers to reach their activity goals and possible solutions to tackle these barriers. During the other four website visits, participants receive feedback about their behavior change process and their action plan (did they reach their goal)? During these website visits, they can adapt their action plans.
  Arms: Intervention group

SUMMARY:
The beneficial effects of physical activity (PA) for older adults are well known. Yet, few older adults reach the health guideline of 150 minutes/week of moderate-intensity PA. eHealth interventions are effective in raising PA levels in older adults on the short-term. However, intermediate- or long-term effects have been examined rarely. This study aimed to investigate the effect of the eHealth intervention 'MyPlan 2.0' on both accelerometer-based and self-reported PA levels in Belgian older adults on the short- and intermediate-term.

This study was a randomized controlled trial with three measurement moments (baseline (n=72), post (five weeks after baseline; n=68) and follow-up (three months after baseline; n=68). At all measurement moments, participants in the control group and intervention group filled out the International Physical Activity Questionnaire and wore an accelerometer during one week. Participants in the intervention group got access to the eHealth intervention 'MyPlan 2.0' and used it for five consecutive weeks after baseline. 'MyPlan 2.0' was based on self-regulatory theory and focused on both pre- and post-intentional processes to increase PA.

DETAILED DESCRIPTION:
Technical information about the content of the MyPlan 2.0. intervention:

MyPlan 2.0. was the eHealth intervention that was used in this study. MyPlan 2.0. is a theory- and user-based intervention. Theories used to develop the intervention are the self-regulation theory and the Health Action Approach model. The intervention targets pre- and post-intentional processes to reach behavior change. The intervention consists of five website visits in five weeks (one per week).

During the first website visit, the participants fill in a short PA questionnaire and based on the answers, they receive personal feedback about their behavior (pre-intentional processes). Knowledge is also provided by giving users the chance to fill in an optional quiz about PA and its beneficial effects. Post-intentional processes are targeted during this first visit by asking the participants to make an action plan. Participants are asked what they want to do (e.g. being more active by cycling during leisure time), when (e.g. every Sunday morning), where (e.g. in the streets nearby) and for how long (e.g. 60 minutes). After answering these questions, the participants can identify difficult situations and possible barriers (i.e. coping planning) while pursuing their goals. Dependent on which barriers they select, specific solutions are given and the participants could choose which ones they consider appropriate and want to apply. After this first website visit, the users can indicate how they want to self-monitor their behaviour (e.g. using an agenda).

One week after finishing the first website visit, the participants receive an email to revisit the website. During this second visit, they receive feedback about their behavioural change process and their goals (e.g. did the participant reach his/her goal or not?). Afterwards the participants have the possibility to adapt their action plan (e.g. setting new, more realistic goals). They can reconsider coping plans, based on barriers they experienced while pursuing their goals. Furthermore, participants can optionally read activity tips. Website visits 3, 4 and 5 are respectively activated one week after the previous visit. Again, the participants are reminded by email. These three last visits are identical to the second visit (review of the action and coping plan).

ELIGIBILITY:
Inclusion Criteria:

* retired
* able to walk 100 meters without assistance
* speak and understand Dutch
* have an email address

Exclusion Criteria:

* severe physical health problems
* not retired
* not able to speak and understand Dutch
* not having an email address

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
change in accelerometer-based physical activity | change between baseline and post (5 weeks after baseline)
  participants wear an accelerometer (activity monitor) to objectively measure their physical activity levels. The investigators examine change in total physical activity (sum of light- intensity and moderate-to-vigorous physical activity) and moderate-to-vigorous physical activity. Higher values represent more physical activity.
change in accelerometer-based physical activity | change between baseline and follow-up (3 months after baseline)
  participants wear an accelerometer (activity monitor) to objectively measure their physical activity levels. The investigators examine change in total physical activity (sum of light-intensity and moderate-to-vigorous physical activity) and moderate-to-vigorous physical activity.
change in self-reported physical activity | change between baseline and post (5 weeks after baseline)
  the validated International Physical Activity Questionnaire (IPAQ) is used to assess self-reported weekly physical activity in three domains (leisure-time, transport, household). Within each domain, different intensities and types of physical activity are assessed. Minutes per week of physical activity in all subdomains are assessed, namely leisure-time walking, leisure-time moderate physical activity, leisure-time vigorous physical activity, moderate physical activity in the garden, vigorous physical activity in the garden, moderate physical activity at home, walking for transport and cycling for transport. The physical activity data are truncated to realistic maxima based on the official IPAQ guidelines. These guidelines subscribe that the maximum amount of physical activity for each subdomain is maximum 840 minutes per week.
change in self-reported physical activity | change between baseline and follow-up (3 months after baseline)
  the validated International Physical Activity Questionnaire (IPAQ) is used to assess self-reported weekly physical activity in three domains (leisure-time, transport, household). Within each domain, different types and intensities of physical activity are assessed. Minutes per week of physical activity in all subdomains are assessed, namely leisure-time walking, leisure-time moderate physical activity, leisure-time vigorous physical activity, moderate physical activity in the garden, vigorous physical activity in the garden, moderate physical activity at home, walking for transport and cycling for transport. The physical activity data are truncated to realistic maxima based on the official IPAQ guidelines. These guidelines subscribe that the maximum amount of physical activity for each subdomain is maximum 840 minutes per week.

CONTACTS AND LOCATIONS:
Overall Officials: Greet Cardon, PhD, Principal Investigator — University Ghent

IPD SHARING:
Plan to Share IPD: Yes
only researchers of our own research group will have access to the full data of the participants, only for research purposes. Only anonymized data will be shared with other researchers of our own research group.
  other researchers can obtain research information upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the data will be available when the study is finished (June 2017) and will be available for ten years.
Access Criteria: the data will be stored on the Ghent University share system that can be accessed with a personal log in and password

REFERENCES:
- [Derived] Van Dyck D, Herman K, Poppe L, Crombez G, De Bourdeaudhuij I, Gheysen F. Results of MyPlan 2.0 on Physical Activity in Older Belgian Adults: Randomized Controlled Trial. J Med Internet Res. 2019 Oct 7;21(10):e13219. doi: 10.2196/13219. PMID 31593541